CLINICAL TRIAL: NCT02718404
Title: 3 Tesla Magnetic Resonance Guided High Intensity Focused Ultrasound (MR-HIFU) in the Treatment of Pain From Bone Metastases of Solid Tumors
Brief Title: 3 Tesla Magnetic Resonance Guided High Intensity Focused Ultrasound in the Treatment of Pain From Bone Metastases of Solid Tumors
Acronym: HIFU-Bone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: following the non-renewal of the loan agreement for the medical device
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST198.01
Record Dates: First submitted 2016-01-21; First posted 2016-03-24 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-05

CONDITIONS: Solid Tumors
Keywords: MR-HIFU; bone metastases; pain treatment
MeSH Terms: conditions — Agnosia | interventions — Dosage Forms; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR-HIFU Treatment (Experimental): The Philips MR-HIFU Sonalleve System integrates a high intensity phased array focused ultrasound transducer with a 3 Tesla Magnetic Resonance (MR) imaging system and electromechanical transducer positioning system to deliver spatially and temporally controlled ultrasound energy and thermal heat to tissues non-invasively.
  At HIFU day (day 0) before treatment patient will be performed a bone lesion MRI and a functional brain MRI.
  During the treatment procedure, an intravenous catheter will deliver MR contrast media and medications (such as sedation and analgesics if required) within the MR room.
  Following the MR-HIFU procedure, a set of MR images of the target region will be acquired with the use of a MR contrast agent, together with a functional brain MRI.
  Interventions: Procedure: MR-HIFU Treatment; Drug: MR contrast media and medications; Procedure: MR images

INTERVENTIONS:
Procedure: MR-HIFU Treatment — The Philips MR-HIFU Sonalleve System integrates a high intensity phased array focused ultrasound transducer with a 3 Tesla Magnetic Resonance (MR) imaging system and electromechanical transducer positioning system to deliver spatially and temporally controlled ultrasound energy and thermal heat to tissues non-invasively.
  At HIFU day (day 0) before treatment patient will be performed a bone lesion MRI and a functional brain MRI.
Drug: MR contrast media and medications — During the treatment procedure, an intravenous catheter will deliver MR contrast media and medications (such as sedation and analgesics if required) within the MR room.
  Other Names: sedation; analgesics
Procedure: MR images — Following the MR-HIFU procedure, a set of MR images of the target region will be acquired with the use of a MR contrast agent, together with a functional brain MRI.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Philips Sonalleve 3 Tesla MR-HIFU device for treating painful bone metastases.

DETAILED DESCRIPTION:
This study is a single centre, single arm, non-randomized, non-blinded study. All eligible subjects will receive MR-HIFU therapy, and no blinding is necessary.

All patients will receive one session of MR-HIFU treatment with the Philips Sonalleve MR-HIFU device on the most painful of their bone metastases.

Will be enrolled in the study consecutive patients with painful skeletal metastases from any solid tumours. Patients with all severity grade of pain (mild, moderate and severe pain) will be included in the study.

At HIFU day (day 0) before treatment patient will be performed a bone lesion MRI and a functional brain MRI. The functional brain MRI is not clinical practice: it is not dangerous for the patient, it only involves a longer time of exam for the patient in the MRI site.

A Brief Pain Inventory, a EORTC-quality of life questionnaire-C15-paired-associate learning and information about pain medication recording will be collected always before treatment.

During the treatment procedure, an intravenous catheter will deliver MR contrast media and medications (such as sedation and analgesics if required) within the MR room. The body temperature of the patients will be measured prior to the procedure. In the MR room the patients will lie still on the HIFU patient table inside the MRI magnet. The operator will locate the target tissue and mark the volume to be treated using MRI images. The operator starts the treatment and monitors the progress of the treatment with MR thermal and dose maps according to the Sonalleve Instructions for Use to ensure safety. Following the MR-HIFU procedure, a set of MR images of the target region will be acquired with the use of a MR contrast agent, together with a functional brain MRI. The functional brain MRI is not clinical practice: it is not dangerous for the patient, it only involves a longer time of exam for the patient under the MRI tunnel. Patients will return for follow-up appointments on Day 14, 30, 60 and 90 for clinical examination. Clinical examination will include inspection and palpation of the treated area and assessment of functionality (e.g. walking pattern or range of movement). The Brief Pain Inventory and the EORTC-quality of life questionnaire will also be administered (to be completed by the patient), and pain medication usage and any possible adverse events will be recorded. Additionally, bone MRI of the treated site and functional brain MRI images will be acquired at 30 and 90 days after treatment.

STATISTICAL CONSIDERATIONS To calculate the sample size the optimal two-stage design developed by Simon is used (Richard Simon, Controlled Clinical Trials 1989). Considering a 2 stage study, with a difference p1-p0=20% between a standard treatment (p0=40%) and the investigated treatment (p1=60%) and setting alfa error probability at 0.10 and beta error probability at 0.10, 28 patients will have to be treated in the 1st stage of the trial. If less or equal than 11 responses are observed among the 28 patients, then the study will be stopped. Otherwise the study will continue to a total of 41 patients will be treated in the second stage. If there are more than 20 responses in 41 patients in the second stage, this treatment could be considered active.

The Intent-to-treat (ITT) population is defined as the population of all enrolled patients. The per-protocol population is considered as all patients in the ITT population except those who prove non to be eligible after enrollment, who withdraw before the MR-HIFU treatment or who commit major protocol violations. The safety population as considered as all patients in the ITT population who underwent to MR-HIFU treatment.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic evidence of bone metastases (BM) from any solid tumors in patients with age ≥ 18 years
* Patient capable of giving informed consent and able to attend study visits
* All target lesion (s) at intended treatment site accessible for MR-HIFU Distance Skin-lesion (target) > 1 cm
* Patient has 1-3 painful lesions, and only the most painful lesion will be treated
* Weight < 140 Kg
* Intended target volume visible by non-contrast MRI
* Patient able to characterize pain at site of target lesion (s), before and after the procedure.
* MR-HIFU treatment date ≥ 2 weeks from last local treatment of the target lesion

Exclusion Criteria:

* Planned treatment lesion is a primary bone tumor Patient enrolled in another clinical study related to bone metastases treatment or pain relief treatment
* Unable to tolerate required stationary position during treatment
* Need for surgical stabilization in case of (impending) fracture (lytic lesion in weight-bearing bone larger than 50% of bone diameter)
* Pregnant woman
* Pain related to target lesion is predominantly due to fracture or impending fracture
* Pain related to target lesion is due to involvement of a neighboring major nerve by the metastatic tumor (cord or nerve compression)
* Target < 3cm from bladder / bowel / nerve along the beam path and < 1cm in the plane orthogonal to the beam
* Target in contact with hollow viscera
* Target located in skull, joints, ribs (when HIFU beam overlapping with lung), spine (excluding sacrum which is allowed) or sternum.
* Scar along proposed HIFU beam path
* Internal or external fixation device along the proposed HIFU beam path or at the target
* MRI contraindicated (e.g. paramagnetic implants, pacemaker, claustrophobia)
* MRI contrast agent contraindicated (e.g. previous anaphylaxis or glomerular filtration rate < 30 ml/min/1.73m2)
* Sedation contraindicated
* Clinically relevant medical history or abnormal physical findings that could interfere with the safety of the participant as judged by the treating physician or investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Pain response | up to 90 days after study treatment
  multidimensional score: the Brief Pain Inventory

SECONDARY OUTCOMES:
Time to pain palliation | up to 30 days after study treatment
  calculated as time from MR-HIFU to pain palliation (achievement of CR or PR)
Time to pain progression | up to 30 days after study treatment
  calculated as time from MR-HIFU to pain progression.
Duration of pain palliation | up to 30 days after study treatment
  calculated as time from pain palliation to pain progression.
Recording of pain medication | 24 hours before study treament
  As proxy measure of "Ongoing or background pain" will be assumed the "present pain intensity"
Quality of Life on the EORTC-QLQ-C15-PAL scale12 | 0, 3, 7, 14 and 30 days following treatment, and additionally at 60 and at 90 days if the subject has not been referred to an alternative local treatment
  measured on the EORTC-QLQ-C15-PAL scale12
Local Tumor Control | at 30 days and 90 days after study treatment
  reduction of metastatic lesion, number of patients with partial or complete response at 30 and 90 days according to MD Anderson criteria and PERCIST criteria.
Side effects | up to 90 days after study treatment
  Incidence of adverse events
  • Incidence of treatment-related adverse events: i. device-related adverse events (resulting from MR-HIFU treatment) ii. study-related adverse events (resulting from protocol-specific procedures)
reduction/increase of tumor markers | at day 14, 30 and 90 after study treatment
  relation to pain relief and local tumor control at the same timepoints repect to the baseline levels.
identification of the brain regions involved in oncological pain | up to 90 days after study treatment
  involved in oncological pain at rest, and the contrast between the brain regions activated before and after the MR-HIFU procedure, related to perceived pain.

CONTACTS AND LOCATIONS:
Overall Officials: Toni Ibrahim, MD, Study Chair — IRST IRCCS
Locations (1):
- Centro di Osteoncologia e Tumori Rari (CDO-TR) IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) S.r.l, Meldola, FC, Italy